CLINICAL TRIAL: NCT03538951
Title: Phase 2B Open-Label Study to Evaluate the Efficacy, Safety, and Tolerability of Topical VDA-1102 Ointment in Subjects With Actinic Keratosis
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Topical VDA-1102 Ointment in Subjects With Actinic Keratosis
Acronym: Phase2b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vidac Pharma (Industry)
Collaborators: Therapeutics, Inc. (Industry); PharPoint Research, Inc. (Industry); Medistat Ltd., Israel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VDA-CP-05
Record Dates: First submitted 2018-04-29; First posted 2018-05-29 (Actual); Results first posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2021-05

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; efficacy; safety; VDA-1102
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: 3-part, open-label, multi-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 10% VDA-1102
  Interventions: Drug: 10% VDA-1102
- Cohort 2 (Experimental): 20% VDA-1102
  Interventions: Drug: 20% VDA-1102

INTERVENTIONS:
Drug: 10% VDA-1102 — 200 mg twice-daily for 12 weeks
  Other Names: 10% VDA-1102 topical ointment
  Arms: Cohort 1
Drug: 20% VDA-1102 — 200 mg once-daily for 12 weeks
  Other Names: 20% VDA-1102 topical ointment
  Arms: Cohort 2

SUMMARY:
This is a Phase 2 clinical study in patients with actinic keratosis involving daily application of 1 of 2 strengths of VDA-1102 topical ointment for approximately 12 weeks (84 days). This study has no placebo and the subjects enrolled in the study will know exactly what they are receiving. The objectives of the study are to evaluate the safety and benefit of these two strengths.

DETAILED DESCRIPTION:
This Phase 2 clinical trial is a 3-part, open-label, multi-center study involving a non-occluded, daily topical dermal application of 1 of 2 strengths of VDA-1102 ointment for approximately 12 weeks (84 days) to an initial 2 cohorts of subjects. The first 40 eligible subjects will be enrolled into Cohort 1 (Part A). Cohort 1 subjects will be assigned to receive approximately 200 mg of 10% VDA-1102 twice-daily (BID). Once approximately 40 subjects have been enrolled in Cohort 1, Cohort 1 will be closed to enrollment and Cohort 2 (Part B) will be opened for enrollment. Cohort 2 subjects will be assigned to receive approximately 200 mg of 20% VDA-1102 once-daily (QD). Once approximately 40 subjects have been enrolled in Cohort 2, an additional 70 subjects will be randomly assigned to Cohort 1 or Cohort 2 (Part C) in a 1:1 ratio.

To qualify for the study, subjects aged 18 (inclusive) or older must have signed informed consent and met the study enrollment criteria that include having 4-8 actinic keratosis (AK) lesions within an approximate 25 cm2 area on the cheek, forehead, or hairless scalp (the "Treatment Field").

ELIGIBILITY:
Inclusion Criteria:

* 4-8 grade 1 or grade 2 AK lesions in Treatment Field on face or scalp

Exclusion Criteria:

* Subject has no clinically significant findings at Baseline
* Subject is unable to demonstrate adequate precision applying the study drug to the Treatment Field at Baseline
* Subject has in the opinion of the Investigator (a) an unstable medical, psychiatric, social problem
* Subject has at any time been given a diagnosis or treatment associated with immunosuppression
* Subject has received VDA-1102 in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Therapeutics Clinical Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 41 | 42
Completed | 40 | 40
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (7.5) | 66.4 (9.2) | 66.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 35 | 33 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 41 | 42 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 42 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance Rate
Description: Efficacy will be evaluated by the proportion of subjects achieving complete clearance of AK lesions in the treatment field of subjects in each treatment arm
Time Frame: Week 16
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 40
Participants | 7 | 9

2. Primary Outcome: Complete Facial Clearance Rate
Description: Efficacy will be evaluated by the proportion of subjects achieving complete clearance of facial AK lesions in the treatment field of subjects in each treatment arm
Time Frame: Week 16
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 26 | 29
Participants | 5 | 8

3. Secondary Outcome: Partial Clearance
Description: Efficacy will be evaluated by the proportion of subjects achieving at least 75% clearance of AK lesions in the selected area of subjects of subjects in each treatment arm
Time Frame: 16 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 40
Participants | 12 | 14

4. Secondary Outcome: Partial Facial Clearance
Description: Efficacy will be evaluated by the proportion of subjects achieving at least 75% clearance of facial AK lesions in the selected area of subjects in each treatment arm
Time Frame: 16 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 26 | 29
Participants | 8 | 13

5. Secondary Outcome: Lesion Number Reduction
Description: Efficacy will be evaluated by the proportion of AK lesion reduction in the treatment field of subjects in each treatment arm
Time Frame: 16 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 40
percentage of change from baseline | -46.00 (36.47) | -52.66 (37.31)

6. Secondary Outcome: Lesion Number Reduction on Face
Description: Efficacy will be evaluated by the proportion of AK lesion reduction in the facial treatment fields of subjects in each treatment arm
Time Frame: 16 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 26 | 29
Percentage of change from baseline | -48.51 (37.35) | -62.42 (34.02)

7. Post Hoc Outcome: Complete Clearance in Patients With Local Skin Reaction- Erythema
Description: Erythema (score=0 or score >0) week 8 100% clearance week 16 (Face and Scalp)
Time Frame: Week 16
Population: Data analyzed by patients with erythema score =0 or > 0
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 40 | 39
Participants
  Erythema score = 0: number analyzed (Participants) | 23 | 28
  Erythema score = 0: Complete clearance | 2 | 4
  Erythema score = 0: No complete clearance | 21 | 24
  Erythema score > 0: number analyzed (Participants) | 17 | 11
  Erythema score > 0: Complete clearance | 5 | 6
  Erythema score > 0: No complete clearance | 12 | 5

8. Post Hoc Outcome: Lesion Reduction in Patients With Local Skin Reaction- Erythema
Description: Erythema (score=0 or score >0) week 8 75% clearance week 16 (Face and Scalp)
Time Frame: Week 16
Population: Data no analyzed for cohort 1 (10% VDA-1102)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 37
Participants
  Erythema score=0: number analyzed (Participants) | 0 | 28
  Erythema score=0: 75% lesion reduction | 0 | 5
  Erythema score=0: Less than 75% lesion reduction | 0 | 23
  Erythema score >0: number analyzed (Participants) | 0 | 9
  Erythema score >0: 75% lesion reduction | 0 | 6
  Erythema score >0: Less than 75% lesion reduction | 0 | 3

ADVERSE EVENTS:
Time Frame: From screening until week 16
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 10/41 | 10/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=41) | Cohort 2 (N=42)
Skin reaction (Skin and subcutaneous tissue disorders) | 10 (14) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03538951/Prot_SAP_000.pdf